CLINICAL TRIAL: NCT00813514
Title: Does VEGF or Complement Factor H Gene Polymorphism Play a Role in the Treatment Success With VEGF Inhibitors in Patients With CNV?
Brief Title: Does Vascular Endothelial Growth Factor (VEGF) or Complement Factor H Gene Polymorphism Play a Role in the Treatment Success With VEGF Inhibitors in Patients With Choroidal NeoVascularization (CNV)?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Fuchsjäger- Mayrl, Department of Clinical Pharmacology, Medical University Vienna, Austria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-270907
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Choroidal NeoVascularization; Age-Related Macular Degeneration
Keywords: AMD; VEGF genotyping; complement H gene polymorphism; Vascular Endothelial Growth Factor A
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration

ARMS (1):
- 1 (Experimental): Open longitudinal study with observer masked analysis
  Interventions: Genetic: VEGF genotyping

INTERVENTIONS:
Genetic: VEGF genotyping — blood sample for gene analysis

SUMMARY:
Age related macular degeneration (AMD) is a multifactorial disease with a strong genetic component. Most importantly a genetic polymorphism in the gene encoding for the complement factor H (CFH) has been recently identified which is highly associated with an increased risk of developing AMD. This Tyr402His polymorphism located on chromosome 1q31 has been implicated to play a role in the development of the disease.

For this purpose a total of 200 patients with wet AMD will be included in the study. As described in detail below, the current study aims to identify potentially non-responders to anti-VEGF therapy based on genetic analysis of VEGF polymorphism and complement factor H polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 50 years
* Angiographically verified neovascular AMD
* Active primary or recurrent subfoveal lesion with CNV secondary to AMD
* Activity to be proven by fluorescein angiography
* Best corrected visual acuity assessed using ETDRS charts of 20/40 to 20/320 in the study eye
* CNV to be treated with intravitreal ranibizumab
* Signed informed consent

Exclusion Criteria:

* Prior treatment with any intravitreal drug in the study eye
* Prior treatment with verteporfin photodynamic therapy in the study eye
* Prior treatment with systemic bevacizumab
* Prior treatment with any intravitreal drug or verteporfin photodynamic therapy in the non-study eye within the 3 moths before the study entry
* Laser photocoagulation within 1 month before study entry in the study eye
* Previous participation in any clinical trial within 1 month before the entry of the study
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either of the two eye due to causes other than AMD such as histoplasmosis or pathological myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye that could either require medical or surgical intervention during the 12 month study period or that could contribute to a loss of best corrected visual acuity over the 12 months study period (e.g. diabetic retinopathy, cataract, uncontrolled glaucoma). The decision on exclusion is to be based on the opinion of the local principal investigator.
* Active intraocular inflammation
* Acute angle-closure glaucoma or narrow angle glaucoma due to the risk of IOP elevation caused by the administration of tropicamide

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual acuity using ETDRS charts | 2 x 5 minutes
Central retinal thickness (Optical coherence tomography) | 2 x 20 minutes
VEGF genotyping | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Leopold Schmetterer, Prof. Dr., Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria